CLINICAL TRIAL: NCT04569786
Title: A Phase 1, Randomized, Double-Blind, Placebo-Controlled, Dose-Ranging Trial to Evaluate the Safety and Immunogenicity of V590 in Healthy Adults
Brief Title: Dose Ranging Trial to Assess Safety and Immunogenicity of V590 (COVID-19 Vaccine) in Healthy Adults (V590-001)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The study was terminated based on an interim assessment of immunogenicity.
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Prevention
Other Study IDs: V590-001; V590-001 (Other: Merck)
Record Dates: First submitted 2020-09-24; First posted 2020-09-30 (Actual); Results first posted 2021-12-29 (Actual); Last update posted 2021-12-29 (Actual); Status verified 2021-12

CONDITIONS: Coronavirus Disease (COVID-19)
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (9):
- V590 5.00x10^5 pfu (Panel A) (Experimental): Participants in this 18 to 54-year-old SARS-CoV-2 seronegative cohort (Panel A) will receive a single dose of V590 5.00x10^5 pfu or placebo on Day 1.
  Interventions: Biological: V590; Other: Placebo
- V590 2.40x10^6 pfu (Panel B) (Experimental): Participants in this 18 to 54-year-old SARS-CoV-2 seronegative cohort (Panel B) will receive a single dose of 2.40x10^6 pfu or placebo on Day 1.
  Interventions: Biological: V590; Other: Placebo
- V590 1.15x10^7 pfu (Panel C) (Experimental): Participants in this 18 to 54-year-old SARS-CoV-2 seronegative cohort (Panel C) will receive a single dose of 1.15x10^7 pfu or placebo on Day 1.
  Interventions: Biological: V590; Other: Placebo
- V590 5.55x10^7 pfu (Panel D) (Experimental): Participants in this 18 to 54-year-old SARS-CoV-2 seronegative cohort (Panel D) will receive a single dose of V590 5.55x10^7 pfu or placebo on Day 1.
  Interventions: Biological: V590; Other: Placebo
- Part 2: 5.00x10^5 pfu (Panel E) (Experimental): Participants in this ≥ 55 years old SARS CoV-2 seronegative cohort (Panel E) will receive a single dose of V590 5.00x10^5 pfu or placebo on Day 1.
  Interventions: Biological: V590; Other: Placebo
- Part 2: 2.40x10^6 pfu (Panel F) (Experimental): Participants in this ≥ 55 years old SARS-CoV-2 seronegative cohort (Panel F) will receive a single dose of 2.40x10^6 pfu or placebo on Day 1.
  Interventions: Biological: V590; Other: Placebo
- Part 2: 1.15x10^7 pfu (Panel G) (Experimental): Participants in this ≥ 55 years old SARS-CoV-2 seronegative cohort (Panel G) will receive a single dose of V590 1.15x10^7 pfu or placebo on Day 1
  Interventions: Biological: V590; Other: Placebo
- Part 2: 5.55x10^7 pfu (Panel H) (Experimental): Participants in this ≥ 55 years old SARS-CoV-2 seronegative cohort (Panel H) will receive a single dose of V590 5.55x10^7 pfu or placebo on Day 1.
  Interventions: Biological: V590; Other: Placebo
- Part 3: 5.55x10^7 pfu (Panel I) (Experimental): Participants in this 18 to 54-year-old SARS-CoV-2 seropositive cohort (Panel I) will receive a single dose of V590 5.55x10^7 pfu or placebo on Day 1.
  Interventions: Biological: V590; Other: Placebo

INTERVENTIONS:
Biological: V590 — Single dose of V590 administered via intramuscular (IM) injection with dosage levels of 5.00x10^5 pfu/mL (Panels A, E), 2.40x10^6 pfu/mL (Panels B,F), 1.15x10^7 pfu/mL (Panels C, G), 5.55x10^7 pfu/mL (Panels D, H, I).
Other: Placebo — Placebo administered via IM injection.

SUMMARY:
The primary objective of this study is to evaluate the safety and tolerability of V590 versus placebo and to assess the immunogenicity of V590 on Day 28. The primary hypothesis is that at least one well-tolerated dose of V590 increases the geometric mean titers (GMTs) of anti-severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) spike serum neutralizing antibody, as measured by plaque reduction neutralization test (PRNT), compared to placebo.

DETAILED DESCRIPTION:
This study was terminated and study objectives, endpoints, and procedures were modified accordingly via Protocol Amendment 03. Analysis included the intervention doses (V590 5.00 x 10^5 plaque forming units [pfu], V590 2.4 x 10^6 pfu, V590 1.15 x 10^7 pfu, V590 5.55 x 10^7 pfu or placebo) as specified in the protocol.

ELIGIBILITY:
Inclusion Criteria:

* Is in overall good health based on medical history, physical examination, and vital sign (VS) measurements performed prior to randomization, as assessed by the investigator.
* Is in overall good health based on laboratory safety tests obtained at the screening visit.
* Has a body mass index (BMI) ≤30 kg/m2 inclusive (after rounding to the nearest whole number).
* Parts 1 and 2 (Panels A-H) only: Has negative testing for severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) based on both antibody and reverse transcription polymerase chain reaction (RT-PCR), at screening and upon start of domiciling.
* Part 3 (Panel I) only: Has positive serology (antibody) testing for SARS-CoV-2, also with negative SARS CoV-2 RT-PCR testing at screening and upon start of domiciling, and without symptoms of respiratory infection for at minimum 3 weeks preceding screening.
* Has been practicing social distancing for at least two weeks prior to planned start of domiciling and has had no close contacts with known active SARS-CoV-2 infection in that time period.
* Is male or female, from 18 years to 54 years of age inclusive (Parts 1 and 3 [Panels A-D, I]) or ≥ 55 years of age (Part 2 [Panels E-H]) at the time of signing the informed consent.
* Male participants are eligible to participate if they agree to the following during the intervention period and for at least 2 months after administration of study intervention: be abstinent from heterosexual intercourse as their preferred and usual lifestyle and agree to remain abstinent OR agree to use contraception unless confirmed to be azoospermic (vasectomized or secondary to medical cause).
* A female participant is eligible to participate if she is not pregnant or breastfeeding, and at least one of the following conditions applies: is not a woman of childbearing potential (WOCBP), or is a WOCBP and using an acceptable contraceptive method, or is abstinent from heterosexual intercourse as their preferred and usual lifestyle. A WOCBP must have a negative highly sensitive pregnancy test before the first dose of study intervention. If a urine test cannot be confirmed as negative, a serum pregnancy test is required.

Exclusion Criteria:

* Has a known hypersensitivity to any component of V590 or placebo.
* Has any known or suspected active clinically significant autoimmune disease or immunosuppressive condition, acquired or congenital, as determined by medical history and/or physical examination.
* Has thrombocytopenia or other coagulation disorder contraindicating intramuscular vaccination or repeated venipuncture.
* Has history or current evidence of any condition, therapy, laboratory abnormality, or other circumstance that might expose the participant to risk by participating in the study, confound the results of the study or interfere with the participant's participation for the full duration of the study.
* Has a history of ongoing liver disease or, at the time of screening, has any one of the following: Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) > 1.5 × Upper Limit of Normal (ULN), alkaline phosphatase and direct bilirubin > ULN (total bilirubin may be up to 2 × ULN as long as direct bilirubin is equal to or below the ULN), or prothrombin time (PT) international normalized ratio (INR) > 1.25.
* Has a history of asthma or allergic asthma that required systemic corticosteroids in the previous year.
* Has a history of Guillain-Barré syndrome.
* Has a history of diabetes mellitus, requiring medication at the time of assessment, OR has a hemoglobin A1c ≥ 6.5.
* Has a history of any medical condition that would put the participant at risk for severe SARS-CoV-2 disease as judged by the investigator.
* Has any ongoing, symptomatic, acute or chronic illness requiring medical or surgical care or any condition that is immunosuppressive.
* Is mentally or legally incapacitated, has significant emotional problems at the time of screening visit or expected during the conduct of the study or has a history of clinically significant psychiatric disorder of the last 5 years.
* Has a history of cancer (malignancy).
* Participant has an estimated glomerular filtration rate (eGFR) ≤60 mL/min/1.73 m^2.
* Has a history of significant multiple and/or severe allergies or has had an anaphylactic reaction or significant intolerability to a vaccine or prescription or non-prescription drugs or food as judged by the investigator.
* Is positive for hepatitis B surface antigen, hepatitis C antibodies or human immunodeficiency virus (HIV)-1 or 2 antibodies. Individuals with antibodies to hepatitis C may be enrolled if hepatitis C viral load is negative and there is no evidence of or history of liver disease.
* Had major surgery, donated or lost 1 unit of blood (approximately 500 mL) within 4 weeks prior to the pre-study (screening) visit.
* A WOCBP who has a positive urine or serum pregnancy test before vaccination.
* A WOCBP who is breastfeeding.
* Has any unstable chronic medical condition, including one that has resulted in change in therapy (medication or other) in the 30 days prior to randomization or hospitalization in the previous year or might be predicted to result in hospitalization in the year after enrollment.
* Has received or is expected to receive any SARS-CoV-2 vaccine or other coronavirus vaccine during the study (except V590), is using investigational agents for prophylaxis of SARS-CoV-2 or is taking any systemic antiviral medications.
* Has received any intra-articular steroid injections within the 3 months prior to study vaccination or is expected to require intra-articular steroid injection during the study.
* Is receiving immunosuppressive therapy or has received immunosuppressive therapy within 6 months of enrollment.
* Has received a blood transfusion or blood products, including immunoglobulin, in the 3 months before anticipated study vaccination.
* Is expected to be receiving or is currently receiving antipyretic or analgesic medication on a daily or every other day basis from randomization through Day 7
* Has ever participated in an investigational study of a SARS-CoV-2 vaccine, a coronavirus vaccine, or an antiviral or other biologic product intended for the treatment of COVID-19.
* Has participated in another vaccine study within 3 months prior to screening or has participated in an investigational study within 4 weeks prior to the screening visit.
* Has ever received a vaccine based on vesicular stomatitis virus (VSV).
* Has a Fridericia's corrected time from Q wave to T wave (QTcF) interval >470 msec (male) or >480 msec (female), has a history of risk factors for Torsades de Pointes, or has uncorrected hypokalemia or hypomagnesemia.
* Is under the age of legal consent.
* Is smoking or vaping and/or has a history of chronic smoking or vaping within approximately six months prior to planned vaccination.
* Does not agree to follow the alcohol restrictions
* Has a tattoo, scar, or other physical finding at the area of the vaccination site that would interfere with intramuscular injection or a local tolerability assessment.
* Is a regular user of any illicit drugs or has a history of drug (including alcohol) abuse within approximately 1 year.
* Presents any concern by the investigator regarding safe participation in the study or for any other reason the investigator considers the participant inappropriate for participation in the study.
* Lives in a nursing home or long-term care facility.
* Is currently working in an occupation with high risk of exposure to SARS-CoV-2 (e.g., health care worker with direct patient contact, emergency response personnel).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 232 (Actual)
Dates: Start 2020-10-29 (Actual); Primary Completion 2021-02-18 (Actual); Study Completion 2021-02-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (7):
- United States (7):
  - Celerion ( Site 0002), Tempe, Arizona
  - Clinical Pharmacology of Miami ( Site 0003), Miami, Florida
  - QPS Miami Research Associates ( Site 0005), South Miami, Florida
  - Bio-Kinetic Clinical Applications (QPS) ( Site 0006), Springfield, Missouri
  - Celerion ( Site 0001), Lincoln, Nebraska
  - Alliance for Multispecialty Reseach, LLC ( Site 0004), Knoxville, Tennessee
  - Worldwide Clinical Trials ( Site 0007), San Antonio, Texas

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Derived] Robbins JA, Tait D, Huang Q, Dubey S, Crumley T, Cote J, Luk J, Sachs JR, Rutkowski K, Park H, Schwab R, Howitt WJ, Rondon JC, Hernandez-Illas M, O'Reilly T, Smith W, Simon J, Hardalo C, Zhao X, Wnek R, Cope A, Lai E, Annunziato P, Guris D, Stoch SA. Safety and immunogenicity of intramuscular, single-dose V590 (rVSV-SARS-CoV-2 Vaccine) in healthy adults: Results from a phase 1 randomised, double-blind, placebo-controlled, dose-ranging trial. EBioMedicine. 2022 Aug;82:104138. doi: 10.1016/j.ebiom.2022.104138. Epub 2022 Jul 6. PMID 35809371
- [Derived] Kreuzberger N, Hirsch C, Chai KL, Tomlinson E, Khosravi Z, Popp M, Neidhardt M, Piechotta V, Salomon S, Valk SJ, Monsef I, Schmaderer C, Wood EM, So-Osman C, Roberts DJ, McQuilten Z, Estcourt LJ, Skoetz N. SARS-CoV-2-neutralising monoclonal antibodies for treatment of COVID-19. Cochrane Database Syst Rev. 2021 Sep 2;9(9):CD013825. doi: 10.1002/14651858.CD013825.pub2. PMID 34473343

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The planned enrollment total was approximately 252 participants.
Groups:
- V590 5.00x10^5 Plaque Forming Units (Pfu): Participants received a single dose of V590 5.00x10^5 pfu on Day 1.
- V590 2.40x10^6 Pfu: Participants received a single dose of V590 2.40x10^6 pfu on Day 1.
- V590 1.15x10^7 Pfu: Participants received a single dose of V590 1.15x10^7 pfu on Day 1.
- V590 5.55x10^7 Pfu: Participants received a single dose of V590 5.55x10^7 pfu on Day 1.
- Placebo: Participants received single dose placebo administered via intramuscular (IM) injection on Day 1.
Period: Overall Study
Arm/Group | V590 5.00x10^5 Plaque Forming Units (Pfu) | V590 2.40x10^6 Pfu | V590 1.15x10^7 Pfu | V590 5.55x10^7 Pfu | Placebo
Started | 39 | 39 | 42 | 56 | 56
Completed | 38 | 39 | 38 | 49 | 55
Not Completed | 1 | 0 | 4 | 7 | 1
Not completed — Lost to Follow-up | 1 | 0 | 4 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 5 | 1
Not completed — Physician Decision | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | V590 5.00x10^5 Plaque Forming Units (Pfu) | V590 2.40x10^6 Pfu | V590 1.15x10^7 Pfu | V590 5.55x10^7 Pfu | Placebo | Total
Number analyzed (Participants) | 39 | 39 | 42 | 56 | 56 | 232
Age, Continuous [Mean (Standard Deviation); unit: Years] | 48.9 (18.8) | 50.9 (16.0) | 51.0 (13.7) | 48.0 (16.1) | 47.3 (16.9) | 49.0 (16.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 22 | 23 | 32 | 29 | 118
  Male | 27 | 17 | 19 | 24 | 27 | 114
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 13 | 20 | 13 | 31 | 19 | 96
  Not Hispanic or Latino | 26 | 19 | 29 | 25 | 37 | 136
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 1 | 0 | 2
  Asian | 0 | 1 | 1 | 0 | 2 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 3 | 5 | 4 | 7 | 8 | 27
  White | 35 | 33 | 35 | 48 | 46 | 197
  More than one race | 0 | 0 | 2 | 0 | 0 | 2
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With at Least 1 Solicited Injection Site Adverse Event
Description: An adverse event (AE) is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study intervention. Solicited injection site AEs (injection site redness/erythema, pain, swelling) were assessed.
Time Frame: Up to 5 days post-vaccination
Population: The analysis population consisted of all randomized participants who received at least one dose of study vaccination.
Measure: Number; unit: Percentage of Participants
Arm/Group | V590 5.00x10^5 Plaque Forming Units (Pfu) | V590 2.40x10^6 Pfu | V590 1.15x10^7 Pfu | V590 5.55x10^7 Pfu | Placebo
Number analyzed (Participants) | 39 | 39 | 42 | 56 | 56
Percentage of Participants
  Injection site redness/erythema | 0.0 | 0.0 | 0.0 | 1.8 | 0.0
  Injection site pain | 28.2 | 35.9 | 31.0 | 42.9 | 46.4
  Injection site swelling | 0.0 | 2.6 | 2.4 | 3.6 | 0.0

2. Primary Outcome: Percentage of Participants With at Least 1 Solicited Systemic Adverse Event
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study intervention. Solicited systemic AEs (joint stiffness/arthralgia, tiredness/fatigue, headache, joint swelling, muscle pain/myalgia, nausea, oral disorder, and rash) were assessed.
Time Frame: Up to 28 days post-vaccination
Population: The analysis population consisted of all randomized participants who received at least one dose of study vaccination.
Measure: Number; unit: Percentage of Participants
Arm/Group | V590 5.00x10^5 Plaque Forming Units (Pfu) | V590 2.40x10^6 Pfu | V590 1.15x10^7 Pfu | V590 5.55x10^7 Pfu | Placebo
Number analyzed (Participants) | 39 | 39 | 42 | 56 | 56
Percentage of Participants
  Joint stiffness/arthralgia | 5.1 | 7.7 | 0.0 | 12.5 | 8.9
  Tiredness/fatigue | 10.3 | 15.4 | 11.9 | 12.5 | 16.1
  Headache | 15.4 | 12.8 | 9.5 | 16.1 | 19.6
  Joint swelling | 0.0 | 0.0 | 0.0 | 1.8 | 3.6
  Muscle pain/myalgia | 10.3 | 7.7 | 0.0 | 10.7 | 7.1
  Nausea | 5.1 | 5.1 | 0.0 | 3.6 | 8.9
  Oral disorder | 0.0 | 0.0 | 0.0 | 1.8 | 1.8
  Rash | 10.3 | 0.0 | 2.4 | 3.6 | 0.0

3. Primary Outcome: Percentage of Participants With at Least 1 Unsolicited Adverse Event
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study intervention. Participants with reported unsolicited AEs were assessed.
Time Frame: Up to ~28 days post-vaccination
Population: The analysis population consisted of all randomized participants who received at least one dose of study vaccination.
Measure: Number; unit: Percentage of Participants
Arm/Group | V590 5.00x10^5 Plaque Forming Units (Pfu) | V590 2.40x10^6 Pfu | V590 1.15x10^7 Pfu | V590 5.55x10^7 Pfu | Placebo
Number analyzed (Participants) | 39 | 39 | 42 | 56 | 56
Percentage of Participants | 6 | 10 | 13 | 21 | 16

4. Primary Outcome: Percentage of Participants With at Least 1 Medically Attended Adverse Event
Description: A medically attended adverse event (MAAE) is an AE in which medical attention is received during an unscheduled, non-routine outpatient visit, such as an emergency room visit, office visit, or an urgent care visit with any medical personnel for any reason. Any MAAE was assessed.
Time Frame: Up to 28 days post-vaccination
Population: The analysis population consisted of all randomized participants who received at least one dose of study vaccination.
Measure: Number; unit: Percentage of Participants
Arm/Group | V590 5.00x10^5 Plaque Forming Units (Pfu) | V590 2.40x10^6 Pfu | V590 1.15x10^7 Pfu | V590 5.55x10^7 Pfu | Placebo
Number analyzed (Participants) | 39 | 39 | 42 | 56 | 56
Percentage of Participants | 0.0 | 0.0 | 0.0 | 5.4 | 0.0

5. Primary Outcome: Percentage of Participants With at Least 1 Serious Adverse Event
Description: A serious adverse event (SAE) is "life threatening," requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect or other important medical event. Any SAE was assessed. Active monitoring of SAEs occurred through Day 28 but were collected per protocol till study completion/termination or ~90 days post-vaccination.
Time Frame: Active monitoring through Day 28 post-vaccination (Up to a maximum of ~90 days post-vaccination)
Population: The analysis population consisted of all randomized participants who received at least one dose of study vaccination.
Measure: Number; unit: Percentage of Participants
Arm/Group | V590 5.00x10^5 Plaque Forming Units (Pfu) | V590 2.40x10^6 Pfu | V590 1.15x10^7 Pfu | V590 5.55x10^7 Pfu | Placebo
Number analyzed (Participants) | 39 | 39 | 42 | 56 | 56
Percentage of Participants | 0.0 | 0.0 | 0.0 | 1.8 | 0.0

6. Primary Outcome: Geometric Mean Titers for Serum Neutralizing Antibodies as Measured by Plaque Reduction Neutralization Test
Description: Serum samples were collected and the presence of serum neutralization antibodies (SNAs) were assessed using plaque reduction neutralization test (PRNT). Geometric mean titers (GMTs) and 95% confidence intervals (CIs), GMT ratios and 90% CIs, and p-values are estimated from a longitudinal data analysis (LDA) model and are provided in accordance with the statistical analysis plan.
Time Frame: 28 days post-vaccination
Population: The analysis population consisted of all randomized participants who were seronegative for anti-severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) nucleocapsid antibody through Day 28 with exclusions for important deviations from the protocol that may substantially affect the results of this immunogenicity endpoint.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | V590 5.00x10^5 Plaque Forming Units (Pfu) | V590 2.40x10^6 Pfu | V590 1.15x10^7 Pfu | V590 5.55x10^7 Pfu | Placebo
Number analyzed (Participants) | 39 | 37 | 41 | 42 | 50
Titer | 6.39 [4.54 to 8.99] | 7.00 [4.93 to 9.92] | 7.67 [5.50 to 10.70] | 15.78 [11.37 to 21.91] | 6.98 [5.17 to 9.42]
Statistical Analysis 1: Comparison: V590 5.00x10^5 Plaque Forming Units (Pfu) vs Placebo; Test type: Superiority — A conclusion of superiority is based on the lower limit of the 90% CI for the estimated GMT ratio (V590/Placebo) being >1.0 (one-sided p-value <0.05); p = 0.649, Longitudinal data analysis (LDA) method — 1-sided; GMT ratios and 90% CIs, and p-values are estimated from an LDA model and are provided in accordance with the statistical analysis plan; GMT Ratio = 0.92, 90% CI 2-sided [0.63 to 1.34]
Statistical Analysis 2: Comparison: V590 2.40x10^6 Pfu vs Placebo; Test type: Superiority — [test comment as in outcome 6, analysis 1]; p = 0.495, LDA model — 1-sided; [statistical method as in outcome 6, analysis 1]; GMT Ratio = 1.00, 90% CI [0.68 to 1.48]
Statistical Analysis 3: Comparison: V590 1.15x10^7 Pfu vs Placebo; Test type: Superiority — [test comment as in outcome 6, analysis 1]; p = 0.339, LDA Model — 1-sided; [statistical method as in outcome 6, analysis 1]; GMT Ratio = 1.10, 90% CI 2-sided [0.75 to 1.60]
Statistical Analysis 4: Comparison: V590 5.55x10^7 Pfu vs Placebo; Test type: Superiority — [test comment as in outcome 6, analysis 1]; p < 0.001, LDA Model — 1-sided; [statistical method as in outcome 6, analysis 1]; GMT Ratio = 2.26, 90% CI 2-sided [1.56 to 3.28]

7. Secondary Outcome: Geometric Mean Titers for SNAs as Measured by PRNT- 7 Days
Description: Serum samples were collected and analyzed on a subset of participants but assays were not conducted on all samples that were collected. Due to the early termination of the study, testing was prioritized for the key samples and timepoints that would provide the required safety and immunogenicity data to support programmatic decision-making and subsequent clinical studies. Blank cells indicate that data were not generated and no data were available. The within-group 95% CIs are obtained by exponentiating the CIs of the mean of the natural log values based on the t-distribution.
Time Frame: 7 days post-vaccination
Population: The analysis population consisted of a subset of all randomized participants who received at least one dose of study intervention and had at least 1 result for the analysis endpoint. Due to the early termination of the study, testing was prioritized and data were not generated for all samples and timepoints.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | V590 5.00x10^5 Plaque Forming Units (Pfu) | V590 2.40x10^6 Pfu | V590 1.15x10^7 Pfu | V590 5.55x10^7 Pfu | Placebo
Number analyzed (Participants) | 20 | 7 | 5 | 0 | 7
Titers | 5.32 [4.68 to 6.04] | 17.07 [1.96 to 148.60] | 5.0 [5.0 to 5.0] |  | 9.78 [1.89 to 50.47]

8. Secondary Outcome: Geometric Mean Titers for SNAs as Measured by PRNT- 14 Days
Description: Serum samples were collected for all participants and the presence of SNAs was assessed using PRNT. The within-group 95% CIs are obtained by exponentiating the CIs of the mean of the natural log values based on the t-distribution.
Time Frame: 14 days post vaccination
Population: The analysis population consisted of all randomized participants who were seronegative for anti-SARS-CoV-2 nucleocapsid antibody through Day 14 with exclusions for important deviations from the protocol that may substantially affect the results of this immunogenicity endpoint.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | V590 5.00x10^5 Plaque Forming Units (Pfu) | V590 2.40x10^6 Pfu | V590 1.15x10^7 Pfu | V590 5.55x10^7 Pfu | Placebo
Number analyzed (Participants) | 39 | 37 | 41 | 42 | 50
Titers | 5.94 [4.66 to 7.56] | 6.64 [4.58 to 9.62] | 7.32 [5.84 to 9.18] | 15.26 [9.73 to 23.95] | 6.45 [4.67 to 8.91]

9. Secondary Outcome: Geometric Mean Titers for Total Anti-Spike Immunoglobulin G Antibodies as Measured by Enzyme-Linked Immunosorbent Assay
Description: Serum samples were collected and the total anti-spike immunoglobulin G (IgG) antibodies were assessed using enzyme-linked immunosorbent assay (ELISA). The within-group 95% CIs are obtained by exponentiating the CIs of the mean of the natural log values based on the t-distribution.
Time Frame: 7, 14, and 28 days post vaccination
Population: The analysis population consisted of all randomized participants who were seronegative for anti-SARS-CoV-2 nucleocapsid antibody on Days 7, 14 or 28 with exclusions for important deviations from the protocol that may substantially affect the results of this immunogenicity endpoint.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | V590 5.00x10^5 Plaque Forming Units (Pfu) | V590 2.40x10^6 Pfu | V590 1.15x10^7 Pfu | V590 5.55x10^7 Pfu | Placebo
Number analyzed (Participants) | 39 | 39 | 42 | 42 | 52
Titers
  Day 7: number analyzed (Participants) | 39 | 37 | 41 | 42 | 50
  Day 7 | 56.60 [44.04 to 72.75] | 65.78 [43.63 to 99.15] | 51.90 [48.13 to 55.97] | 58.06 [45.70 to 73.77] | 68.36 [47.01 to 99.39]
  Day 14: number analyzed (Participants) | 39 | 37 | 41 | 42 | 50
  Day 14 | 56.01 [44.51 to 70.47] | 65.10 [43.75 to 96.86] | 63.63 [52.31 to 77.39] | 104.12 [72.27 to 150.01] | 67.13 [47.26 to 95.36]
  Day 28: number analyzed (Participants) | 38 | 37 | 40 | 42 | 50
  Day 28 | 62.82 [45.48 to 86.77] | 69.78 [47.31 to 102.93] | 69.14 [53.00 to 90.20] | 107.58 [75.93 to 152.41] | 71.13 [49.82 to 101.57]

10. Secondary Outcome: Number of Participants With Vaccine Viremia as Measured by Reverse Transcription-Polymerase Chain Reaction
Description: Positive viremia was defined as detectable reverse transcription polymerase chain reaction (RT-PCR) results greater than or equal to the lower limit of detection (≥ LLOD); results were deemed quantifiable if the result was greater than or equal to the lower limit of quantification (≥ LLOQ). The number of participants who have a positive V590 RT-PCR result greater than or equal to the lowest limit of detection (≥LLOD) were assessed.
Time Frame: 1, 2, 3, 4, 5, 6, 7, 14 and 28 days post-vaccination
Population: The analysis population consisted of all randomized participants who received study intervention with data available for Days 1, 2, 3, 4, 5, 6, 7, 14, or 28.
Measure: Count of Participants; unit: Participants
Arm/Group | V590 5.00x10^5 Plaque Forming Units (Pfu) | V590 2.40x10^6 Pfu | V590 1.15x10^7 Pfu | V590 5.55x10^7 Pfu | Placebo
Number analyzed (Participants) | 39 | 39 | 42 | 56 | 56
Participants
  Day 1: number analyzed (Participants) | 26 | 20 | 15 | 8 | 22
  Day 1 | 4 | 5 | 9 | 8 | 0
  Day 2: number analyzed (Participants) | 38 | 39 | 42 | 56 | 56
  Day 2 | 6 | 8 | 24 | 54 | 0
  Day 3 | 4 | 5 | 22 | 48 | 0
  Day 4 | 1 | 6 | 9 | 30 | 0
  Day 5: number analyzed (Participants) | 22 | 17 | 14 | 6 | 19
  Day 5 | 1 | 0 | 0 | 0 | 0
  Day 6: number analyzed (Participants) | 24 | 18 | 16 | 4 | 19
  Day 6 | 0 | 0 | 0 | 0 | 0
  Day 7: number analyzed (Participants) | 28 | 22 | 20 | 36 | 21
  Day 7 | 0 | 0 | 0 | 0 | 0
  Day 14: number analyzed (Participants) | 26 | 15 | 22 | 36 | 16
  Day 14 | 0 | 0 | 0 | 0 | 0
  Day 28: number analyzed (Participants) | 14 | 7 | 19 | 30 | 6
  Day 28 | 0 | 0 | 0 | 0 | 0

11. Secondary Outcome: Number of Participants With Viral Shedding in Saliva as Measured by RT-PCR
Description: The number of participants with viral shedding detected by RT-PCR in saliva specimens was assessed. Only Day 7 samples were assayed for all participants. Day 14 and 28 samples for a participant were assayed if the Day 7 result was positive (≥LLOD). Due to the early termination of the study, testing was prioritized for the key samples and timepoints that would provide the required safety and immunogenicity data to support programmatic decision-making and subsequent clinical studies. Blank cells indicate data were not generated and no data were available. Additional sample testing is not possible because the viral shedding assay is not qualified for samples that have been stored for this length of time.
Time Frame: 1, 2, 3, 4, 5, 6, 7, 14, and 28 days post-vaccination
Population: The analysis population consisted of all randomized participants who received study intervention. Due to the early termination of the study, testing was prioritized and data were not generated for all samples and timepoints.
Measure: Count of Participants; unit: Participants
Arm/Group | V590 5.00x10^5 Plaque Forming Units (Pfu) | V590 2.40x10^6 Pfu | V590 1.15x10^7 Pfu | V590 5.55x10^7 Pfu | Placebo
Number analyzed (Participants) | 39 | 39 | 42 | 56 | 56
Participants
  Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Day 2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Day 3: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Day 4: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Day 5: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Day 6: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Day 7 | 0 | 0 | 0 | 1 | 1
  Day 14: number analyzed (Participants) | 0 | 0 | 0 | 1 | 1
  Day 14 |  |  |  | 0 | 0
  Day 28: number analyzed (Participants) | 0 | 0 | 0 | 1 | 1
  Day 28 |  |  |  | 0 | 0

12. Secondary Outcome: Number of Participants With Viral Shedding in Urine as Measured by RT-PCR
Description: The number of participants with viral shedding detected by RT-PCR in urine specimens was assessed. Due to the early termination of the study, testing was prioritized for the key samples and timepoints that would provide the required safety and immunogenicity data to support programmatic decision-making and subsequent clinical studies. Only Day 7 samples were assayed for all participants. Day 14 and 28 samples for a participant were assayed if the Day 7 result was positive (≥LLOD). Blank cells indicate data were not generated and no data were available.
Time Frame: 1, 2, 3, 4, 5, 6, 7, 14, and 28 days post-vaccination
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | V590 5.00x10^5 Plaque Forming Units (Pfu) | V590 2.40x10^6 Pfu | V590 1.15x10^7 Pfu | V590 5.55x10^7 Pfu | Placebo
Number analyzed (Participants) | 39 | 39 | 42 | 56 | 56
Participants
  Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Day 2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Day 3: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Day 4: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Day 5: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Day 6: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Day 7 | 0 | 0 | 0 | 0 | 0
  Day 14: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Day 28: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

13. Secondary Outcome: Number of Participants With Viral Shedding in Stool (If Assayed) as Measured by RT-PCR
Description: The study was terminated and V590 stool samples for viral shedding (considered optional per protocol) were not assayed. Due to the early termination of the study, testing was prioritized for the key samples and timepoints that would provide the required safety and immunogenicity data to support programmatic decision-making and subsequent clinical studies. Blank cells indicate that data were not generated and no data were available.
Time Frame: 2-4, 5-7 days post-vaccination
Population: The study was terminated based on an interim assessment of immunogenicity and V590 stool samples for viral shedding were not assayed.
Arm/Group | V590 5.00x10^5 Plaque Forming Units (Pfu) | V590 2.40x10^6 Pfu | V590 1.15x10^7 Pfu | V590 5.55x10^7 Pfu | Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Non-serious adverse events were reported up to Day 28 following vaccination. Serious adverse events (SAEs) and the all cause mortality were reported throughout the duration of an individual's study participation (active monitoring through Day 28 post-vaccination [Up to a maximum of ~90 days post-vaccination])
Description: The analysis population consisted of all randomized participants who received at least one dose of study vaccination.
Arm/Group | V590 5.00x10^5 Plaque Forming Units (Pfu) | V590 2.40x10^6 Pfu | V590 1.15x10^7 Pfu | V590 5.55x10^7 Pfu | Placebo
All-Cause Mortality (participants affected / at risk) | 0/39 | 0/39 | 0/42 | 0/56 | 0/56
Serious Adverse Events (participants affected / at risk) | 0/39 | 0/39 | 0/42 | 1/56 | 0/56
Other Adverse Events (participants affected / at risk) | 19/39 | 23/39 | 23/42 | 39/56 | 36/56
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | V590 5.00x10^5 Plaque Forming Units (Pfu) (N=39) | V590 2.40x10^6 Pfu (N=39) | V590 1.15x10^7 Pfu (N=42) | V590 5.55x10^7 Pfu (N=56) | Placebo (N=56)
Amaurosis fugax (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | V590 5.00x10^5 Plaque Forming Units (Pfu) (N=39) | V590 2.40x10^6 Pfu (N=39) | V590 1.15x10^7 Pfu (N=42) | V590 5.55x10^7 Pfu (N=56) | Placebo (N=56)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lymphocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ear discomfort (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Asthenopia (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal tenderness (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (2) | 1 (1) | 1 (2) | 2 (3) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 2 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Eructation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal sounds abnormal (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lip swelling (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (4) | 2 (2) | 0 (0) | 2 (3) | 5 (7)
Oral disorder (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Tongue disorder (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chest discomfort (General disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 0 (0)
Fatigue (General disorders) | 4 (8) | 6 (7) | 5 (6) | 7 (13) | 9 (13)
Feeling cold (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Feeling hot (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypothermia (General disorders) | 0 (0) | 1 (4) | 0 (0) | 1 (1) | 0 (0)
Injection site bruising (General disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Injection site erythema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Injection site haemorrhage (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Injection site induration (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Injection site movement impairment (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Injection site pain (General disorders) | 11 (13) | 14 (16) | 13 (14) | 24 (28) | 27 (35)
Injection site swelling (General disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Injection site warmth (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Malaise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Peripheral swelling (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Asymptomatic COVID-19 (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Urethritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lip injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Muscle strain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Scratch (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin laceration (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood fibrinogen increased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Liver function test increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
SARS-CoV-2 antibody test positive (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (3) | 3 (3) | 0 (0) | 7 (8) | 5 (7)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 4 (4) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 2 (2)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 4 (5) | 3 (5) | 0 (0) | 6 (9) | 4 (7)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Ageusia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anosmia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 6 (6) | 5 (8) | 4 (4) | 9 (17) | 11 (20)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Poor quality sleep (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Fear (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lower respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (2)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 4 (4) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Flushing (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hot flush (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
The study was terminated based on an interim assessment of immunogenicity.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If publication activity is not directed by the Sponsor, the investigator agrees to submit all manuscripts or abstracts to the Sponsor before submission. This allows the Sponsor to protect proprietary information and to provide comments. Authorship will be determined by mutual agreement and in line with International Committee of Medical Journal Editors authorship requirements.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-02-17): https://cdn.clinicaltrials.gov/large-docs/86/NCT04569786/Prot_SAP_000.pdf